CLINICAL TRIAL: NCT03895255
Title: Randomized Non-inferiority Trial of Selective Splenic Flexure Mobilization for the Formation of Low Colorectal Anastomosis After Total Mesorectal Excision and D3 Paraaortic Lymph Node Dissection in Low Rectal Cancer.
Brief Title: Selective sPlenic flExure Mobilization for Low colorEctal Anastomosis After D3 lYmph Node Dissection (Speedy Trial)
Acronym: SpeeDy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683472
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Rectal Cancer
Keywords: lymph node dissection; high tie; low tie; splenic flexure mobilization; anastomotic leak
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMA high ligation with routine SFM (Active Comparator): Inferior mesenteric artery is ligated close to its origin. Splenic flexure is always mobilized.
  Interventions: Procedure: Paraaortic lymph node dissection, IMA high ligation, TME, routine splenic flexure mobilization
- IMA skeletonization and low ligation with selective SFM (Experimental): Inferior mesenteric artery is ligated below the origin of left colic artery. Splenic flexure is mobilized only if needed.
  Interventions: Procedure: Paraaortic lymph node dissection, IMA low ligation, TME, selective splenic flexure mobilization

INTERVENTIONS:
Procedure: Paraaortic lymph node dissection, IMA high ligation, TME, routine splenic flexure mobilization — Nerve-sparing paraaortic lymph node dissection is performed. The inferior mesenteric artery is divided at 1-2 cm from its origin from the aorta. Nerve-sparing total mesorectal excision is performed. Splenic flexure is mobilized. Side-to-end sigmoido-rectal anastomosis is created.
  Other Names: High tie with routine SFM
  Arms: IMA high ligation with routine SFM
Procedure: Paraaortic lymph node dissection, IMA low ligation, TME, selective splenic flexure mobilization — Nerve-sparing paraaortic lymph node dissection is performed. Then inferior mesenteric artery is skeletonized down to the origin of left colic artery and divided below it. Nerve-sparing total mesorectal excision is performed. Splenic flexure is mobilized only if sigmoid colon is unsuitable for anastomosis or doesn't reach the rectal stump. Then descending-rectal side-to-end anastomosis is created.
  Other Names: Low tie with selective SFM
  Arms: IMA skeletonization and low ligation with selective SFM

SUMMARY:
In the Low Anterior Resection of rectum for cancer, the section level of IMA and the need of SFM is still debated.

The aim of this study is to explore the different impacts of high and low ligation with peeling off vascular sheath of inferior mesenteric artery (IMA) in low anterior resection of the rectum for cancer. This study purpose to demonstrate that low IMA ligation, sparing of left colic artery (LCA) and selective SFM results in higher anastomotic leakage rate than high IMA ligation with routine SFM (with the difference of more than 5%).

DETAILED DESCRIPTION:
Although TME is the standard curative operation for rectal cancer patients, who undergo low anterior resection (LAR) or abdominoperineal resection (APR) with a permanent colostomy, the strategy to restore the transit between colon and rectum (in case of LAR) is still debated in literature.

Several studies comparing high-tie with low-tie ligation reported a stage-specific survival benefit for high-tie, but on the other hand recent studies demonstrated that low-tie, without splenic flexure mobilization (SFM), decreases the complexity of the laparoscopic procedure and could reduces the operating time with comparable oncological outcomes.

The method of restorative surgery, after Total Mesorectal Excision (TME), largely depends on the length of the resected part of the colon, that is related to patient's anatomical features and the height of vascular ligation performed during the operation.

In attempt to perform a radical paraaortic lymph node dissection the inferior mesenteric artery (IMA) is usually ligated at its origin and the Arcade of Riolan provides bloody supply to any distal anastomosis. Unfortunately the Arcade of Riolan is an inconstant finding and sometimes (26% of cases) is mandatory to mobilize the splenic flexure to ensure a safe and tension-free anastomosis. SFM is a time-consuming component of LAR, has the additional risk of iatrogenic splenic injury and is very difficult during a laparoscopic resection.

In 2005 was demonstrated that routine SFM is not always necessary during anterior resection for rectal cancer.

A recent retrospective analysis by Mouw showed that SFM was associated with wider margins and a decreased rate of inadequate nodal staging in patients undergoing LAR.

This trial aims to demonstrate that low IMA ligation, sparing of LCA and selective SFM results in higher anastomotic leakage rate than high IMA ligation with routine SFM (with the difference of more than 5%). Furthermore this study purpose to evaluate the need to perform splenic flexure mobilization (SFM) in low ligation group and the, operation time, apical lymph nodes positive rate and short terms postoperative complication in both groups

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary rectal adenocarcinoma located within 15 cm from anal verge not involving internal and/or external sphincter muscle
2. Stage I-III
3. Elective surgical treatment with TME and primary colorectal anastomosis
4. Receive or not receive neoadjuvant radio-chemotherapy
5. Overall health status according to American Society of Anesthesiologists (ASA) classification: I-III
6. Signed informed consent with agreement to attend all study visits
7. The patient is not pregnant

Exclusion Criteria:

1. Unresectable tumour, inability to perform a TME with colorectal anastomosis, inability to complete R0 resection or presence of T4b tumour necessitating a multi-organ resection
2. The patient wants to withdraw from the clinical trial
3. Loss to follow-up
4. Inability to complete all the trial procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2016-10-02 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2021-11-02 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage Rate | 4-6 weeks
  The rate of symptomatic and asymptomatic colorectal anastomotic leakage

SECONDARY OUTCOMES:
Operating time | 1 day
  The duration of surgical procedure
Intraoperative complications rate | 1 day
  The rate of complications during surgery
Splenic flexure mobilization rate | 1 day
  The rate of splenic flexure mobilization in Low tie group
Conversion rate | 1 day
  The rate of conversion from laparoscopic or robotic approach to open approach
IMA architectonics | 1 day
  The incidence of left colic artery, first, second and third sigmoid arteries
The length of IMA trunk | 1 day
  the length of inferior mesenteric artery trunk based on preoperative CT-scans and intraoperative findings
Early postoperative complications rate | 30 days
  The rate of complications in first 30 days after surgery
Specimen morphometry | 30 days
  The gross dimensions of resected specimen: length, the distal and proximal resection margins distance, vascular pedicle length
Positive Apical Lymph Nodes Rate | 30 days
  The rate of metastatic lymph nodes found in the area of paraaortic lymph node dissection
Complications of defunctioning stoma | 3 month
  Any complications of defunctioning stoma
The postoperative hospital stay | 1 month
  the number of days from the first day after operation to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery, Moscow, Russia

REFERENCES:
- [Result] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Result] Ho YH. Techniques for restoring bowel continuity and function after rectal cancer surgery. World J Gastroenterol. 2006 Oct 21;12(39):6252-60. doi: 10.3748/wjg.v12.i39.6252. PMID 17072945
- [Result] Kanemitsu Y, Hirai T, Komori K, Kato T. Survival benefit of high ligation of the inferior mesenteric artery in sigmoid colon or rectal cancer surgery. Br J Surg. 2006 May;93(5):609-15. doi: 10.1002/bjs.5327. PMID 16607682
- [Result] Lange MM, Buunen M, van de Velde CJ, Lange JF. Level of arterial ligation in rectal cancer surgery: low tie preferred over high tie. A review. Dis Colon Rectum. 2008 Jul;51(7):1139-45. doi: 10.1007/s10350-008-9328-y. Epub 2008 May 16. PMID 18483828
- [Result] Mouw TJ, King C, Ashcraft JH, Valentino JD, DiPasco PJ, Al-Kasspooles M. Routine splenic flexure mobilization may increase compliance with pathological quality metrics in patients undergoing low anterior resection. Colorectal Dis. 2019 Jan;21(1):23-29. doi: 10.1111/codi.14404. Epub 2018 Sep 29. PMID 30184316
- [Result] Katory M, Tang CL, Koh WL, Fook-Chong SM, Loi TT, Ooi BS, Ho KS, Eu KW. A 6-year review of surgical morbidity and oncological outcome after high anterior resection for colorectal malignancy with and without splenic flexure mobilization. Colorectal Dis. 2008 Feb;10(2):165-9. doi: 10.1111/j.1463-1318.2007.01265.x. Epub 2007 May 16. PMID 17506796